CLINICAL TRIAL: NCT04708405
Title: The Relationship Between Helicobacter Pylori Infection and Inflammatory Bowel Diseases: A Real-life Observation
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Collaborators: High Institute of Public Health, Egypt (Other)
Responsible Party: Principal Investigator, Ekram Abdel Wahab, Assistant professor, Alexandria University
Other Study IDs: 622-2019
Record Dates: First submitted 2021-01-06; First posted 2021-01-14 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Inflammatory Bowel Diseases; Helicobacter Pylori Infection
Keywords: Inflammatory Bowel Diseases; Helicobacter Pylori; Egypt
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inflammatory bowel disease patients: Inflammatory bowel disease patients screened for Helicobacter Pylori Infection
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Follow up and observe under standard of care given

SUMMARY:
Numerous epidemiological studies have investigated the association between Helicobacter pylori (H. pylori) infection and inflammatory bowel disease (IBD) with various conflicting results. The main objective of this study is to further explore the possible association between H. pylori infection and IBD and its impact on disease course. The investigators sought to conduct a prospective observational study and enroll a total of 182 IBD patients who were screened for H. pylori infection. All the participants will be clinically evaluated at the initial visit and bimonthly for 3 months. Several factors will be explored such are diet, physical activity, life style and considering specific environmental exposures that impact the development of disease or its relapse.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with inflammatory bowel disease condition

Exclusion Criteria:

* Having irritable bowel disease
* Being younger than 18 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients diagnosed with inflammatory bowel disease condition
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Change in the inflammatory bowel disease condition | 3 months
  Change in the inflammatory bowel disease condition during follow up as measured by disease related symptoms [weight loss where weight will be measured and reported in kilograms]
Change in the inflammatory bowel disease condition | 3 months
  Change in the inflammatory bowel disease condition during follow up as measured by frequency of disease related symptoms [number of attacks disease related symptoms per day (diarrhea, tenesmus, bleeding per rectum, abdominal pain, indigestion)]
Change in the inflammatory bowel disease condition | 3 months
  Change in the inflammatory bowel disease condition during follow up as measured by changes in baseline laboratory parameters measured in serum samples [C reactive protein (IU/ml)]
Change in the inflammatory bowel disease condition | 3 months
  Change in the inflammatory bowel disease condition during follow up as measured by changes in baseline laboratory parameters measured in serum samples [Hemoglobin (g/dl)]
Change in the inflammatory bowel disease condition | 3 months
  Change in the inflammatory bowel disease condition during follow up as measured by changes in baseline laboratory parameters measured in blood samples [Complete blood picture including white blood count per cmm, platelets count per cmm]
Change in the inflammatory bowel disease condition | 3 months
  Change in the inflammatory bowel disease condition during follow up as measured by changes in baseline laboratory parameters measured in serum samples [ESR (mm/hr)]
Change in the inflammatory bowel disease condition | 3 months
  Change in the inflammatory bowel disease condition during follow up as measured by changes in baseline laboratory parameters measured in serum samples [Fasting blood glucose (mg/dl)]

CONTACTS AND LOCATIONS:
Locations (1):
- High Institute of Public Health, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
publication